CLINICAL TRIAL: NCT07385443
Title: Creación de un Nodo Integral Para la Distrofia Miotónica Tipo 1 en España: Registro clínico, Mapas genómicos, epigenómicos y proteómicos (DM1-Hub)
Brief Title: The Spanish National Registry for Myotonic Dystrophy Type 1
Acronym: DM1-Hub
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: Instituto de Investigacion Sanitaria INCLIVA (Other); Biobizkaia (Unknown); Biogipuzkoa Health Research Institute (Other); Germans Trias i Pujol Hospital (Other); Hospital Infanta Sofia (Other); Hospital de Basurto (Other); Hospital Donostia (Other); Hospital Universitario Virgen del Rocio (Unknown); Hospital Universitario Marqués de Valdecilla (Other); Complejo Hospitalario Universitario de Albacete (Other); Hospital Universitario La Fe (Other); Hospital Univeritario Ntra. Sra. de la Candelaria (Unknown)
Responsible Party: Sponsor
Other Study IDs: PMPER24/00007
Record Dates: First submitted 2025-12-31; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Myotonic Dystrophy 1; DM1; Myotonic Dystrophy Type 1; Myotonic Dystrophy, Congenital; Steinert Disease
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — DNA samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myotonic Dystrophy Type 1 (DM1): The group included Individuals with a confirmed genetic diagnosis of Myotonic Dystrophy Type 1 (DM1)
  Interventions: Other: Patient Registry
- Control: The group included control subjects as individuals without a genetic diagnosis of Myotonic Dystrophy Type 1 (DM1).
  Interventions: Other: Patient Registry

INTERVENTIONS:
Other: Patient Registry — Patient Registry

SUMMARY:
Myotonic Dystrophy Type 1 (DM1) is a rare genetic neuromuscular condition that can affect multiple organs and varies widely in how it presents. DM1 is the most common form of adult-onset muscular dystrophy, with an estimated prevalence of approximately 1-5 per 10,000 people. In Spain, the condition shows notable regional differences, making it especially important to understand its characteristics within the population.

The aim of this study is to support a research initiative designed to better characterise DM1. We are developing a comprehensive national registry, collecting patient-reported information, clinical data and omics data that will improve our understanding of the disease and help identify individuals who may be eligible for clinical trials.

DETAILED DESCRIPTION:
The DM1-Hub Patient Registry (https://www.dm1spain.com/) aims to recruit individuals living in Spain with a confirmed genetic diagnosis of myotonic dystrophy type 1 (DM1). Participants may be referred by healthcare professionals or patient organizations. They may also learn about the registry through outreach activities, informational materials, collaborations with national and local patient associations, DM1-Hub events, or through their own online searches.

After completing the informed consent process with their neurologist, participants are connected with the DM1-Hub patient support staff assigned to their hospital. An appointment is scheduled, and all the data collected is entered into the REDCap database.

The objective of this study is to establish a Natural History Patient Registry for individuals with DM1 in Spain. Participants will be invited to take part in follow-up assessments to support the characterization of disease progression over time. A parallel control group will also be recruited to facilitate biomarker discovery and improve understanding of factors associated with disease prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Myotonic Dystrophy Type 1 (DM1) through genetic testing.

Exclusion Criteria:

* There are no exclusion criteria for the registry

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with Myotonic Dystrophy Type 1 (DM1) will volunteer to participate in this study. The study will be advertised through physician recommendations, outreach and educational activities directed at neuromuscular professionals, the registry website, national and local patient associations, and through patient-focused events, conferences, and scientific meetings across Spain.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Genomic Caracterization | 1 year, year 1
  Long-read genomic sequencing analyses encompassing CTG expansion characterization and whole-genome genetic and epigenetic profiling.

SECONDARY OUTCOMES:
Proteomic Characterization | 1 year, year 1
  Biomarker evaluation
WAIS IV neuropsychological tests | 2 years, year 1
  IQ, memory, attention, language
vHOT | 1 year, year 1
  Video Hand Opening Time, clinical measure for Myotonic Dystrophy (DM1) tracking hand reopening speed
Muscular Impairment Rating Scale (MIRS) | 1 year, year 1
  The Muscular Impairment Rating Scale is a 5-point ordinal clinical scale used to evaluate the severity of muscular impairment in patients with myotonic dystrophy.
  Scores range from 1 (minimal or no impairment) to 5 (severe muscle impairment). Higher scores indicate worse functional impairment.
Hand Grip Strength | 1 year, year 1
  Hand grip strength is assessed as a measure of upper limb muscle strength using a hand-held dynamometer. Grip strength is measured separately in the dominant and non-dominant hand, and recorded in kilograms (kg).
  For each hand, three consecutive attempts are performed, alternating between hands to minimize fatigue. The maximum value (best of three attempts) for each hand is recorded and used for analysis.
  Higher values indicate better muscle strength and functional outcome, while lower values reflect greater muscular impairment.
6MWT | 1 year, year 1
  Six-Minute Walk Test
10MWRT | 1 year, year 1
  10-meter Walk/Run Test
30CST | 1 year, year 1
  30-Second Chair Stand Test
FVC | 1 year, year 1
  Forced Vital Capacity (L)
Electrocardiogram (ECG) | 1 year, year 1
  The following ECG-derived parameters and abnormalities are recorded:
  * PR interval duration (milliseconds)
  * QRS complex duration (milliseconds)
  * Presence of atrioventricular block (AV block) (yes/no), and AV block grade when present (first degree, second degree Mobitz I, second degree Mobitz II, third degree)
  * Presence of supraventricular arrhythmias (yes/no)
  * Presence of ventricular arrhythmias (yes/no)
  * Other electrocardiographic abnormalities, recorded as free text when applicable
  All measurements are extracted from the ECG tracing according to standard clinical practice.
  Higher PR or QRS durations and the presence of conduction abnormalities or arrhythmias indicate greater cardiac involvement, while normal values and absence of abnormalities indicate preserved cardiac electrical function.
BMI | 1 year, year 1
  Body Mass Index
OBGYN events | 1 year, year 1
  Collection of gynecological clinical history and relevant reproductive health events for participants who opt to provide this information.
GI symptomatology | 1 year, year 1
  Collection of participant-reported gastrointestinal symptoms and related clinical information.
MBS (Myotonia Behaviour Scale) | 1 year, year 1
  Myotonia severity is assessed using the Myotonia Behaviour Scale (MBS), a clinician-reported ordinal scale that evaluates the functional impact of myotonia-related muscle stiffness on daily activities.
  The scale ranges from 0 to 5, with higher scores indicating greater severity and functional interference due to myotonia:
  0: No muscle stiffness
  1. Mild stiffness present but easily ignored
  2. Stiffness present and occasionally noticeable but does not interfere with daily activities
  3. Stiffness requiring increased concentration to perform certain tasks or activities
  4. Stiffness interfering with all tasks and daily activities
  5. Severe, disabling stiffness requiring constant movement to avoid complete motor blockage
  Lower scores reflect minimal or absent myotonia, while higher scores reflect greater functional impairment due to myotonia.
Modified Rankin Scale (mRS) | 1 year, year 1
  Global disability is assessed using the Modified Rankin Scale (mRS), a widely used ordinal scale measuring the degree of disability or dependence in daily activities.
  The scale ranges from 0 to 6, with higher scores indicating greater disability or death:
  0: No symptoms
  1. No significant disability; able to carry out all usual activities despite symptoms
  2. Slight disability; unable to perform all previous activities but able to manage own affairs without assistance
  3. Moderate disability; requiring some help but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to bodily needs without help
  5. Severe disability; bedridden, incontinent, and requiring constant nursing care and attention
  6. Death
Patient-Reported Outcome: Quality of life | 1 year, year 1
  INQoL (Individualized Neuromuscular Quality of Life Questionnaire)
Patient-Reported Outcome: Fatigue | 1 year, year 1
  FSS (Fatigue Severity Scale )
Patient-Reported Outcome: Dietary Habits | 1 year, year 1
  MEDAS-14 (Mediterranean Diet Adherence Screener)
Patient-Reported Outcome: Sleepiness | 1 year, year 1
  DSS (Daytime Sleepiness Scale)
Patient-Reported Outcome: Apathy | 1 year, year 1
  AES (Apathy Evaluation Scale)
Patient-Reported Outcome: Physical Activity | 1 year, year 1
  IPAQ (International Physical Activity Questionnaire)
Patient-Reported Outcome: Mental Health | 1 year, year 1
  MHI-5 (Mental Health Inventory)

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Nogales Gadea, Ph.D., Study Director — Germans Trias i Pujol Research Institute; Arturo Lopez Castel, Ph.D., Principal Investigator — INCLIVA Instituto de Investigación Sanitaria; Virginia Arechavala-Gomeza, Ph.D., Principal Investigator — IIS Biobizkaia
Locations (8):
- Spain (8):
  - Hospitals within the DM1 network, Multiple Locations, Andalusia
  - Hospitals within the DM1 network, Multiple Locations, Basque Country
  - Hospitals within the DM1 network, Multiple Locations, Canary Islands
  - Hospitals within the DM1 network, Multiple Locations, Cantabria
  - Hospitals within the DM1 network, Multiple Locations, Castilla-La Macha
  - Hospitals within the DM1 network, Multiple Locations, Catalonia
  - Hospitals within the DM1 network, Multiple Locations, Madrid
  - Hospitals within the DM1 network, Multiple Locations, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: DM1-Hub webpage — https://www.dm1spain.com